CLINICAL TRIAL: NCT00335790
Title: A Prospective, Randomized, Double-Blind, Controlled Study on the Clinical Effects of Hyperbaric Therapy in Autistic Children
Brief Title: A Controlled Trial of the Clinical Effects of Hyperbaric Therapy in Autistic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Hyperbarics Association (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HBA-2
Record Dates: First submitted 2006-06-09; First posted 2006-06-12 (Estimated); Last update posted 2007-04-10 (Estimated); Status verified 2007-04

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Hyperbaric Oxygenation

INTERVENTIONS:
Procedure: Hyperbaric Therapy

SUMMARY:
Autism is a neurodevelopmental disorder currently affecting as many as 1 out of 166 children in the United States. Autism is considered by many to be a permanent condition with little hope for improvement. Treatment for autism is centered on special schooling and behavioral therapy; medical science currently has little to offer. Recent research has discovered that some autistic individuals have decreased blood flow to the brain, evidence of gastrointestinal and brain inflammation, increased markers of oxidative stress, and a relative mitochondrial dysfunction. Hyperbaric oxygen therapy (HBOT) can compensate for decreased blood flow by increasing the oxygen content of plasma and body tissues and can even normalize oxygen levels in ischemic tissue. In addition, animal studies have shown that HBOT has potent anti-inflammatory effects and reduces oxidative stress. Furthermore, recent evidence demonstrates that HBOT increases the production of mitochondria and mobilizes stem cells from human bone marrow, which may aid recovery in neurodegenerative diseases. Based upon these findings, it is hypothesized that HBOT will improve symptoms in autistic individuals.

Our recent retrospective case series demonstrated that HBOT may improve symptoms in autistic children. We recently completed a prospective pilot trial using HBOT in 18 children which demonstrated significant clinical improvements in autistic children on several standardized scales. Most of the scales were parent-rated, although some were rated by teachers. However, parents were not blinded to the fact that their children received HBOT and evaluation of the children was through parent-rated scales, either of which could lead to bias. There was no placebo or control group. Therefore, the improvements found in this prospective study could have been due merely to chance or the natural development of the children. To determine if HBOT improves symptoms in autistic children, a double-blind controlled study is needed.

DETAILED DESCRIPTION:
Autism is a neurodevelopmental disorder currently affecting as many as 1 out of 166 children in the United States. Autism is considered by many to be a permanent, static condition with little hope for improvement. Treatment for autism is centered on special schooling and behavioral therapy; medical science currently has little to offer. Recent research has discovered that some autistic individuals have decreased cerebral perfusion, evidence of gastrointestinal and neuro-inflammation, increased markers of oxidative stress, and a relative mitochondrial dysfunction. Multiple independent single photon emission computed tomography (SPECT) and positron emission tomography (PET) research studies have revealed hypoperfusion to several areas of the autistic brain, most notably the temporal regions and areas specifically related to language comprehension and auditory processing. Several studies show that diminished blood flow to these areas correlates with many of the clinical features associated with autism including repetitive, self-stimulatory and stereotypical behaviors, and impairments in communication, sensory perception, and social interaction. Hyperbaric oxygen therapy (HBOT) has been used with clinical success in several cerebral hypoperfusion syndromes including cerebral palsy, fetal alcohol syndrome, closed head injury, and stroke. HBOT can compensate for decreased blood flow by increasing the oxygen content of plasma and body tissues and can even normalize oxygen levels in ischemic tissue. In addition, animal studies have shown that HBOT has potent anti-inflammatory effects and reduces oxidative stress. Furthermore, recent evidence demonstrates that HBOT increases the production of mitochondria and mobilizes stem cells from human bone marrow, which may aid recovery in neurodegenerative diseases. Based upon these findings, it is hypothesized that HBOT will improve symptoms in autistic individuals.

Our recent retrospective case series demonstrated that HBOT may improve symptoms in autistic children. We recently completed a prospective pilot trial using HBOT in 18 children which demonstrated statistically significant clinical improvements in autistic children on several standardized scales. Most of the scales were parent-rated, although some were rated by teachers. However, parents were not blinded to the fact that their children received HBOT and evaluation of the children was through parent-rated scales, either of which could lead to bias. There was no placebo or control group. Therefore, the improvements found in this prospective study could have been due merely to chance or the natural development of the children. To determine if HBOT improves symptoms in autistic children, a double-blind controlled study is indicated.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of Autistic Disorder, confirmed with Autism Diagnostic Observation Schedule (ADOS) and Autism Diagnostic Interview-Revised (ADI-R)
* HBOT naïve

Exclusion Criteria:

* DSM-IV diagnosis of Pervasive Developmental Disorder other than Autistic Disorder including PDD-NOS (Pervasive Developmental Disorder, not otherwise specified) and Asperger's Syndrome
* Uncontrolled seizures
* Ear infection
* Uncontrolled asthma
* Inability to equalize ear pressure
* Fragile X syndrome
* Current therapy consisting of chelation

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60
Dates: Start 2006-06; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Blinded Therapist Autism Diagnostic Observation Schedule (ADOS)
Blinded Therapist Aberrant Behavior Checklist (ABC-C)
Blinded Physician Clinical Global Impression Severity Score (CGI)
Parental Autism Treatment Evaluation Checklist (ATEC)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Rossignol, MD, Principal Investigator — University of Virginia
Locations (4):
- United States (4):
  - Center for Autism Research and Education, Phoenix, Arizona
  - International Child Development Resource Center, Melbourne, Florida
  - Blue Ridge Spectrum Center, Charlottesville, Virginia
  - Advocates for Children, Lynchburg, Virginia

REFERENCES:
- [Derived] Rossignol DA, Rossignol LW, Smith S, Schneider C, Logerquist S, Usman A, Neubrander J, Madren EM, Hintz G, Grushkin B, Mumper EA. Hyperbaric treatment for children with autism: a multicenter, randomized, double-blind, controlled trial. BMC Pediatr. 2009 Mar 13;9:21. doi: 10.1186/1471-2431-9-21. PMID 19284641